CLINICAL TRIAL: NCT04555759
Title: Validity and Reliability of the 2-minute Walk Test in Individuals With a Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-01473
Record Dates: First submitted 2020-08-26; First posted 2020-09-21 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with spinal cord injuries (Experimental)
  Interventions: Other: 2-minute walk test

INTERVENTIONS:
Other: 2-minute walk test — The patients will do a 2-minute walk test, using their walking aids or braces

SUMMARY:
There exist a variety of outcome measures to asses gait function in individuals with a spinal cord injury (SCI). The most established measures are the 10-meter walk test (10MWT) and the 6-minute walk test (6mWT). They are used to assess treatment efficacy and recovery of gait function in individuals with SCI. However, the 10MWT is appropriate for poor walkers but not sensitive in good walkers and the 6mWT can be time-consuming and is very demanding for severely impaired patients. Therefore the 2-minute walk test (2mWT) has gained more attention in the SCI field. The 2mWT has been established in numerous neurological diseases and has shown to correlate with the 6mWT in patients with neuromuscular disease, multiple sclerosis and stroke. Though the 2mWT has not yet been validated in individuals with SCI.

A limitation that affects all timed walking tests is that they suffer from limited information about gait quality (i.e. how walking function is achieved). Being able to receive information on the gait quality of a patient can help to understand the underlying mechanisms of walking improvements after an intervention (e.g. compensation vs recovery). The research in the field of inertia measuring units (IMU) develops and advances very rapidly at the moment resulting in the possibility to perform a gait analysis with a simple IMU setup. However, the reliability of such measurement setups has not yet been shown in individuals with SCI.

The primary aim of this study is to test the validity and reliability of the 2mWT in the SCI population.

Additionally, it will be investigated if a simple sensor setup can give additional reliable information about the gait pattern of individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling all of the following inclusion criteria are eligible for the study:
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* At least 18 years old
* Spinal cord injury
* Able to walk with a speed of at least 0.17m/s with or without walking devices and or bracing

Exclusion Criteria:

* Current orthopaedic problems of lower limbs
* History of severe cardiac condition
* Premorbid major depression or psychosis
* Unlikely to complete the intervention or return for second visit
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
2-minute walk test (meters an individual walks in 2 minutes) | 1-7 days

SECONDARY OUTCOMES:
Inertia Measuring Unit data | 1-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Armin Curt, Prof., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Schweizer Paraplegiker-Zentrum, Nottwil
  - Balgrist University Hospital, Zurich

REFERENCES:
- [Derived] Willi R, Werner C, Demko L, de Bie R, Filli L, Zorner B, Curt A, Bolliger M. Reliability of patient-specific gait profiles with inertial measurement units during the 2-min walk test in incomplete spinal cord injury. Sci Rep. 2024 Feb 6;14(1):3049. doi: 10.1038/s41598-024-53301-y. PMID 38321085
- [Derived] Willi R, Widmer M, Merz N, Bastiaenen CHG, Zorner B, Bolliger M. Validity and reliability of the 2-minute walk test in individuals with spinal cord injury. Spinal Cord. 2023 Jan;61(1):15-21. doi: 10.1038/s41393-022-00847-1. Epub 2022 Aug 23. PMID 35999254